CLINICAL TRIAL: NCT02227641
Title: Prospective, Open, Randomized, Two-arm, Controlled, Multicenter Clinical Phase I/IIa Trial to Evaluate the Safety and Efficacy of Adoptive Immunotherapy With Allogeneic CMV/EBV Specific, Peptide Stimulated T-cells (CD3+) for Prevention or Preemptive Therapy of Reactivation of CMV and/or EBV in Patients After Allogeneic, HLA Identical Stem Cell Transplantation
Brief Title: Preventative/Preemptive Adoptive Transfer of Peptide Stimulated CMV/EBV Specific T-cells in Patients After Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); University of Regensburg (Other); Johannes Gutenberg University Mainz (Other); Charite University, Berlin, Germany (Other); University Hospital Augsburg (Other); BayImmuNet Bavarian Immunotherapy Network (Unknown); German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: AIT-MULTIVIR-01; 2012-004240-30 (EudraCT Number)
Record Dates: First submitted 2014-08-26; First posted 2014-08-28 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Patients Undergoing Allogeneic Stem Cell Transplantation
Keywords: CMV; Cytomegalovirus; EBV; Epstein Barr Virus; virus; T cell; adoptive transfer; transplantation; allogeneic
MeSH Terms: conditions — Epstein-Barr Virus Infections; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adoptive transfer of CMV/EBV specific T-cells (Experimental): Repetitive adoptive T-cell transfer starting at day 30 after allogeneic stem cell transplantation.
  Interventions: Biological: CMV/EBV specific T-cell
- Control (No Intervention): Observation only.

INTERVENTIONS:
Biological: CMV/EBV specific T-cell — Peptide stimulated allogeneic T-cells with dual specificity for CMV and EBV
  Other Names: T cell
  Arms: Adoptive transfer of CMV/EBV specific T-cells

SUMMARY:
In patients after allogeneic stem cell transplantation reactivation of latent herpesviruses such as Cytomegalovirus (CMV) and Epstein Barr Virus (EBV) is a frequent and life threatening complication requiring antiviral treatment. The underlying problem is a severe suppression of the donors immune system after transplantation into the patient. Herpesviruses such as CMV and EBV persist after primary infection life long in the host and therefore require constant immunological control. This control is largely provided by the T-cell compartment of the immune system. After allogeneic stem cell transplantation the T-cell compartment requires a long time for its reconstitution since only a small fraction of the donor T-cells are transplanted. During this time Herpesviruses can reoccur due to the lack of effective T-cell control.

This study therefore aims at reconstituting the T-cell compartment with CMV and EBV specific T-cells at an early time point after allogeneic stem cell transplantation. It is mainly a phase I study to demonstrate that these in vitro generated T-cells can be applied safely in this patient population. The study also aims at demonstrating the efficacy of CMV/EBV specific T-cells by monitoring viral reactivation and use of antiviral drugs. The hypothesis is, that CMV/EBV specific T-cell can be applied safely and do not result in graft versus host disease and that they successfully prevent reactivation of CMV and EBV after adoptive transfer in patients after allogeneic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Indication for allogeneic stem cell transplantation
* HLA identical donor, related or unrelated, 10/10 match
* Stem cell source: G-SCF mobilized peripheral blood stem cells
* Presence of at least one HLA allele: A0101, A0201, B0702, B0801, B3501, C0702
* Positive EBV serology of the donor
* Positive CMV serology of the donor
* Adequate contraception

Exclusion Criteria:

* Donor CMV seronegative
* Donor EBV seronegative
* Stem cell source: bone marrow or cord blood
* Alemtuzumab for conditioning
* Sorror Score >3
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2016-10 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Toxicity of adoptive transfer of CMV/EBV specific T-cells | 1-28 days after adoptive T-cell transfer
  Assessment of acute transfusion toxicity within 24 hours after adoptive T-cell transfer.
  Assessment of the development of acute transfusion associated acute graft versus host disease (GvHD) within 28 days after adoptive T-cell transfer

SECONDARY OUTCOMES:
Influence of preventative/preemptive adoptive transfer of CMV/EBV specific T-cells on virus reactivation | During observation period until day 204 post transplantation
  Incidence of reactivation of CMV and/or EBV during the observation period assessed by virus specific PCR of peripheral blood.
Influence of preventative/preemptive adoptive transfer of CMV/EBV specific T-cells on the use of antiviral therapy | During observation period until day 204 post transplantation
  Cumulative dose of Ganciclovir, Valganciclovir, Foscarnet, Cidofovir
Influence of preventative/preemptive adoptive transfer of CMV/EBV specific T-cells on the use of Rituximab | During observation period until day 204 post transplantation
  Cumulative dose of Rituximab.
Influence of preventative/preemptive adoptive transfer of CMV/EBV specific T-cells on T-cell reconstitution | During observation period until day 204 post transplantation
  Immunomonitoring of peripheral blood by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Armin H Gerbitz, MD, PhD, Study Director — Charite University, Berlin, Germany; Bernd Spriewald, MD, PhD, Principal Investigator — University Hospital Erlangen; Anita Kremer, MD,PhD, Principal Investigator — University Hospital Erlangen; Katja San Niccolo, MD, Principal Investigator — University Hospital Erlangen
Locations (6):
- Germany (6):
  - Medical Center Augsburg, Augsburg
  - Charité University Hospital Berlin, Berlin
  - Universitiy Hospital Erlangen, Erlangen
  - University of Mainz, Mainz
  - University of Munich LMU, Munich
  - University of Regensburg, Regensburg

REFERENCES:
- [Derived] Gerbitz A, Gary R, Aigner M, Moosmann A, Kremer A, Schmid C, Hirschbuehl K, Wagner E, Hauptrock B, Teschner D, Roesler W, Spriewald B, Tischer J, Moi S, Balzer H, Schaffer S, Bausenwein J, Wagner A, Schmidt F, Brestrich J, Ullrich B, Maas S, Herold S, Strobel J, Zimmermann R, Weisbach V, Hansmann L, Lammoglia-Cobo F, Remberger M, Stelljes M, Ayuk F, Zeiser R, Mackensen A. Prevention of CMV/EBV reactivation by double-specific T cells in patients after allogeneic stem cell transplantation: results from the randomized phase I/IIa MULTIVIR-01 study. Front Immunol. 2023 Oct 30;14:1251593. doi: 10.3389/fimmu.2023.1251593. eCollection 2023. PMID 37965339
- See also: Dept. of Medicine 5, Hematology/Oncology, University of Erlangen — http://www.medizin5.uk-erlangen.de/